CLINICAL TRIAL: NCT06802783
Title: Impact of Procedure Materials on Patient Anxiety, Depression, and Pain in Prostate Biopsy Consent
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MAR.UAD.0017
Record Dates: First submitted 2024-12-23; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Prostate Biopsy
Keywords: prostate biopsy; anxiety; pain; depression
MeSH Terms: conditions — Anxiety Disorders; Pain; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- written consent group (No Intervention): Only traditional written consent will be provided to this group.
- photo-consent group (Active Comparator): Photo consent which show materials use in procedure will be provided to this group before the biopsy
  Interventions: Other: Photo consent

INTERVENTIONS:
Other: Photo consent — The first group was shown photographs of the devices alongside the written consent form, while the second group received only the written consent. The study compared the pain, depression and anxiety scores between the two groups.
  Arms: photo-consent group

SUMMARY:
The gold standard for diagnosing prostate cancer is an ultrasound-guided prostate biopsy. Despite its low complication rates, the procedure can cause significant stress, discomfort and anxiety in patients. This study aimed to determine whether visually introducing the materials (ultrasound, probe, biopsy needle) used during the biopsy could reduce patient anxiety and increase comfort.

DETAILED DESCRIPTION:
Forty patients suspected of having prostate cancer were included in this prospective study. All patients received detailed information about the procedure, but they were divided into two groups. The first group was shown photographs of the devices alongside the written consent form, while the second group received only the written consent. The study compared the pain, depression and anxiety scores between the two groups

ELIGIBILITY:
Inclusion Criteria:

- patient's clinical data indicated the need for a prostate biopsy

Exclusion Criteria:

* included having a diagnosis of psychiatric illness
* having previously undergone a prostate biopsy under local anesthesia
* being a patient under active surveillance for prostate cancer

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety Level | Pre-procedure
  For Anxiety, Hospital Anxiety Scale used. In the Hospital Anxiety Score, the minimum score is 0, and the maximum score is 21. As the score increases, it indicates higher levels of anxiety.
Depression Level | Pre-procedure
  For Depression, Hospital Depression Scale used . In the Hospital Depression Score, the minimum score is 0, and the maximum score is 21. As the score increases, it indicates higher levels of depression.
Pain Level | Pre procedure
  For Pain, Visual Analog Scale used. In the Visual Analog Pain Scale, the minimum score is 0, and the maximum score is 10. As the score increases, it indicates higher levels of pain.

SECONDARY OUTCOMES:
Anxiety Level | Immediately after the procedure
  For Anxiety, Hospital Anxiety Scale used. In the Hospital Anxiety Score, the minimum score is 0, and the maximum score is 21. As the score increases, it indicates higher levels of anxiety.
Depression Level | Immediately after the procedure
  For Depression, Hospital Depression Scale used . In the Hospital Depression Score, the minimum score is 0, and the maximum score is 21. As the score increases, it indicates higher levels of depression
Pain Level | Immediately after the procedure
  For Pain, Visual Analog Scale used. In the Visual Analog Pain Scale, the minimum score is 0, and the maximum score is 10. As the score increases, it indicates higher levels of pain.

CONTACTS AND LOCATIONS:
Overall Officials: BAHADIR SAHIN, Study Director — MARMARA UNİVERSİTY SCHOOL OF MEDİCİNE DEPARTMENT OF UROLOGY
Locations (1):
- Marmara University School of Medicine Urology Department, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No